CLINICAL TRIAL: NCT04800744
Title: Aromatherapy for Improving Post-Surgical Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Beekley Medical (Industry)
Responsible Party: Principal Investigator, Jacques E. Chelly, Professor, Anesthesiology and Perioperative Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY20100091
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Quality of Life; Anxiety Postoperative
Keywords: aromatherapy; unilateral hip replacement surgery; post-surgical quality of life; mastectomy

STUDY DESIGN:
Intervention Model Description: Single-center Prospective, Randomized, Double-blind, Active comparator trial involving patients undergoing unilateral hip replacement and patients undergoing unilateral or bilateral mastectomy that score ≥19 on the PROMIS Emotional Distress - Anxiety - Short Form 8a
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender Peppermint Elequil Aromatab (Experimental): Participants will have a lavender peppermint elequil aromatab applied in same day admissions area at least 1 hour prior to the start of unilateral hip replacement. Thereafter, the participant will apply a new treatment elequil aromatab at 24 hrs, 36 hrs, 48 hrs, and 60 hrs post-operative.
  Interventions: Other: Lavender peppermint elequil aromatab
- Sweet Almond Oil Elequil Aromatab (Active Comparator): Participants will have a sweet almond oil active comparator elequil aromatab applied in same day admissions area at least 1 hour prior to the start of unilateral hip replacement. Thereafter, the participant will apply a new active comparator elequil aromatab at 24 hrs, 36 hrs, 48 hrs, and 60 hrs post-operative.
  Interventions: Other: Sweet almond oil elequil aromatab

INTERVENTIONS:
Other: Lavender peppermint elequil aromatab — Lavender peppermint elequil aromatab applied pre-operatively and every 12 hours thereafter for the duration of the 72 hour treatment window.
  Other Names: treatment aromatab
  Arms: Lavender Peppermint Elequil Aromatab
Other: Sweet almond oil elequil aromatab — Sweet almond oil elequil aromatab applied pre-operatively and every 12 hours thereafter for the duration of the 72 hour treatment window.
  Other Names: active comparator aromatab
  Arms: Sweet Almond Oil Elequil Aromatab

SUMMARY:
Pre-operative anxiety is a very common condition that plagues many patients prior to undergoing surgery. Anxious patients are most frequently treated with sedatives in the perioperative period, which can have a negative impact on post-operative recovery, especially when combined with narcotic pain medications. Pre-operative anxiety, depression and catastrophizing have been shown to be factors leading to an increase of up to 50% of postoperative pain and opioid requirement. Therefore, the control of mood disorders prior to surgery may help with the perioperative pain management and postoperative opioid requirement. The use of essential oils in aromatherapy have long been associated with psychological wellness, and anecdotal reports suggest that aromatherapy, specifically lavender scent, may reduce anxiety. This study will assess the role of the elequil aromatab #373 Lavender-Peppermint in improving post-surgical quality of life in patients undergoing unilateral hip replacement surgery and in patients undergoing unilateral or bilateral mastectomy. Additionally, this study will follow subjects through their perioperative course to measure to what degree the aromatherapy intervention helps to reduce instances of post-operative nausea and vomiting (PONV) and opioid requirement following surgery.

DETAILED DESCRIPTION:
Potential subjects will be recruited from the office of orthopedic surgeon Dr. Michael O'Malley, Dr. Frank Plate or Dr. Brian Klatt, as well as the office of plastic surgeon Dr. Carolyn De La Cruz and will be provided with a recruitment flier. The patient will have the option of contacting our research team to discuss the study further, or, if they express interest in the study to the surgeon's office, their name will be given to us by the surgeon's office staff. If our research team is contacted, or if we reach out based upon the list of interested potential subjects, we will discuss the study over the telephone with the patient with the understanding that they will sign the informed consent with Dr. Chelly or a co-investigator on the day of surgery in the pre-operative area.

Subjects that meet inclusion criteria, self report anxiety, and provide informed consent will complete the PROMIS Emotional Distress - Anxiety - Short Form 8a before completing any other questionnaires. If the subject scores ≥19 on the PROMIS Emotional Distress - Anxiety - Short Form 8a they will be enrolled in the study. However, if the subject scores <19 on the PROMIS Emotional Distress - Anxiety - Short Form 8a they will be considered a screen fail and excluded from participation in the study. Once the subject is enrolled, they will be asked to complete the PROMIS Emotional Distress-Depression-Short Form, the PROMIS Pain Interference - Short Form 6b and the Pain Catastrophizing Scale. After completion of these forms, subjects will be equally randomized to either the active comparator aromatab (sweet almond oil) or treatment aromatab (lavendar peppermint). Study coordinators, Co-Is, and subjects will be blinded.

The aromatab will be placed on the patient's clothing at least one hour prior to surgery while the patient is in same day admission. After surgery, the subject will be assessed for post-operative nausea, pain scores, and pain medication requirement in the PACU and then assessed daily until discharge. At the 12-hour mark, the subject will receive another new patch that is consistent with their randomization arm. They will apply a new patch every 12 hours for the duration of the 72-hour treatment window with the last patch being placed at 60 hrs post-operative.

Upon discharge, subjects will receive patches for the remaining 72-hour treatment window. At this time, subjects will be asked an overall satisfaction questionnaire measured on a scale to 0-10 (0=lowest satisfaction and 10=highest satisfaction).

The subjects will be contacted via Redcap 24 hours, 48 hours and 7 days post-operative and asked to complete PROMIS Emotional Distress - Anxiety - Short Form 8a, the PROMIS Emotional Distress-Depression-Short Form , the PROMIS Pain Interference - Short Form 6b and the Pain Catastrophizing Scale. In addition to this, the subject will be asked to report in a Redcap survey VAS pain score, incidence of nausea and vomiting, and their opioid consumption at 24 hrs, 48 hrs and 7 days post-operative. The subjects will also receive reminders via Redcap at 12hrs, 24hrs, 36hrs, 48hrs, and 60 hrs to change their patch, and will be asked to document in Redcap the time this is complete.

One month following the surgery the subject will be contacted via Redcap to determine their level of pain (VAS), opioid consumption, incidence of nausea and vomiting, functional recovery using SF12, and the PROMIS Emotional Distress - Anxiety - Short Form 8a, the PROMIS Emotional Distress-Depression-Short Form, PROMIS Pain Interference - Short Form 6b and Pain Catastrophizing Scale. Subjects who are contacted via Redcap to complete follow-up questionnaires and do not complete them on the day they are assigned will be contacted via phone for reminder.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and ≤ 80
* Scheduled to undergo unilateral hip replacement surgery or scheduled to undergo unilateral or bilateral mastectomy
* Self-reported anxiety related to upcoming surgery
* Subject is willing and able to provide informed consent
* Subject is willing and able to complete follow-up procedures

Exclusion Criteria:

* Score <19 on the PROMIS Emotional Distress - Anxiety - Short Form 8a
* History of major anxiety or depression
* History of opioid use disorder or alcohol abuse
* History of atrial fibrillation
* History of fibromyalgia
* History of G6PD deficiency
* Plant or tree nut allergy
* Surgery requiring a hospitalization of greater than 3 days
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Change in post-operative anxiety | Day of surgery versus 7 days post-operative
  Demonstrate the effect of the elequil aromatab (Lavender-Peppermint) versus an active comparator (sweet almond oil) on participant's answers to the PROMIS Emotional Distress-Anxiety-Short Form 8a 7 days following surgery. There are 8 questions about how the participants may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.

SECONDARY OUTCOMES:
Post-operative emotional distress related to depression | Day of surgery through one month post-operative
  Post-operative emotional distress related to depression will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Depression-Short Form. There are 8 questions about how the participant many have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Post-operative pain rating using the Visual Analog Scale (VAS) | Day of surgery through one month post-operative
  Post-operative pain ratings will be measured by the assessment of the participant's answers to the Visual Analog Scale (VAS). This measurement is a visual scale from 0-10, with 0 being no pain, 5 being moderate pain and 10 being the worst imaginable pain. The lowest possible score is 0 and the highest possible score is 10.The participant will be asked to score pain at its best and worst over the period since they were last asked. Higher scores present a worse outcome.
Post-operative pain rating using the Pain Catastrophizing Scale | Day of surgery through one month post-operative
  Post-operative pain ratings will be measured by the assessment of the participant's answers to the Pain Catastrophizing Scale questionnaire. There are 13 statements related to pain that participants will record experiencing on a scale of 0 being experienced not at all to 4 being experienced all of the time. The lowest possible score is 0 and the highest possible score is 52. Higher scores present a worse outcome.
Post-operative consequences of pain | Day of surgery through one month post-operative
  Post-operative consequences of pain will be measured by the assessment of the participant's answers to the PROMIS Pain Interference - Short Form 6b. This assessment measures the self-reported consequences of pain on relevant aspects of the participant's physical and social life in the past 7 days. The scale for interference of pain with each activity is from 1, not at all in the past 7 days, to 5, very much in the past 7 days. The overall score can range from 6 to 30. Higher scores present a worse outcome.
Opioid Consumption | Day of surgery through one month post-operative
  Investigate the efficacy of aromatherapy in reducing perioperative opioid consumption in opioid naive subjects undergoing unilateral total hip replacement surgery and those undergoing unilateral or bilateral mastectomy.
Incidence of post-operative nausea and vomiting | Day of surgery through one month post-operative
  Evaluate the incidence of post-operative nausea and vomiting.
Incidence of post-operative complications | Day of surgery through one month post-operative
  Investigate the incidence of post-operative complications in subjects who received the standard protocol for total hip replacement surgery or the standard protocol for mastectomies versus subjects who received the standard protocol and aromatherapy.
Functional Recovery | Day of surgery through one month post-operative
  Functional recovery will be measured by the assessment of the participant's answers to the Functional Recovery Questionnaire 12-Item Short Form Health Survey (SF-12). The SF-12 Health Survey includes questions from the SF-36 Health Survey (Version 1).These include: 2 questions concerning physical functioning; 2 questions on role limitations because of physical health problems; 1 question on bodily pain; 1 question on general health perceptions; 1 question on vitality (energy/fatigue); 1 question on social functioning; 2 questions on role limitations because of emotional problems; and 2 questions on general mental health (psychological distress and well-being). Overall score can range from 12 to 53. Higher scores present a better outcome.
Hospital Readmissions | Day of surgery through one month post-operative
  Determine the number of patients readmitted to the hospital.
Length of Hospital Stay | Day of surgery through one month post-operative
  Evaluate time to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques E Chelly, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No